CLINICAL TRIAL: NCT06871553
Title: The Efficacy of the Self-Management Program on Knowledge and Self-Management Behavior of Hemodialysis Patients at Siem Reap Provincial Referral Hospital, Cambodia
Brief Title: The Self-management Program on Hemodialysis Patients in Cambodia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Responsible Party: Principal Investigator, Hour Sovannara, Principal Investigator, Hiroshima University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 076
Record Dates: First submitted 2025-03-05; First posted 2025-03-12 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Disease on Hemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Self management education program (Experimental): The trained nurses will provide the self-management education program to the patients at the bedside by showing the educational videos and a textbook, at the 1st dialysis session after the intervention period starts.
  The nurses then provide the self-monitoring notebook at the 1st session and teach the patients how to record daily behavior on the notebook. Additionally, the nurses will teach the patients how to properly use various measurement tools, such as a weighing scale, blood pressure machine, water measurement cup, salt measuring spoon, food scale, and urine salt checker for daily monitoring. A measurement cup and a salt measuring spoon will be provided to each patient for free. Majority of patients do not have those tools, the nurses will encourage them to purchase the tools, or the researcher prepares these tools at the dialysis center and let the patients use them at the center. If appropriate, the nurses will rent equipment to patients, if possible.
  Interventions: Other: Self management education program

INTERVENTIONS:
Other: Self management education program — After returning home, patients will be encouraged to practice their self-management behaviors and record the behavior and data to the self-monitoring notebook.
  At their next hemodialysis session, patients will bring their self-monitoring notebook, and the nurse will review the behavior and data, and offering feedback. The nurses will provide additional videos and education, and request the patients to share their experiences with other patients in the hemodialysis room. This cycle of education, self-monitoring, and feedback will continue with each hemodialysis session.

SUMMARY:
Chronic kidney disease (CKD) is a growing global health issue, with increasing numbers of patients requiring kidney replacement therapy (KRT), particularly in low- and middle-income countries. In Cambodia, the prevalence of CKD is rising, and the demand for hemodialysis treatment is straining healthcare resources. This study aims to develop and evaluate the efficacy of a self-management program focused on improving the knowledge and self-management behaviors of hemodialysis patients in Cambodia. This study will use a quasi-experimental pre- and post-design to improve in patients' knowledge and self-management behavior for CKD patients maintaining on hemodialysis at Siem Reap Provincial Referral Hospital, Cambodia from April 2025 to August 2025. The study population consists of patients undergoing hemodialysis in this hospital who meet the following criteria. The sample size was calculated by using the G Power analysis, on the basis effect size of 0.5, an estimated power of 0.8, and of 0.05. A two tailed test was used to calculate that the sample should be 34 patients. However, because of this pilot nature, we include all patients who meet the inclusion criteria (n= 54). The intervention is designed to provide the self-management program to all participant by the trained nurses. Primary outcome: Patients' self-management behavior, as measured by the researcher-developed questionnaire. Secondary outcome include patient' knowledge score, quality of life, self-monitoring (symptoms, blood pressure, weight, diet, fluid intake, exercise, medication), physical and laboratory data (blood pressure, weight, creatinine, urea) and qualitative data (free comments related to their experience and changes of the participation).

DETAILED DESCRIPTION:
In Cambodia, the prevalence of CKD among the adult population is estimated at 1.2% (approximately 0.12 million) and the number of ESKD is unknown. However, in 2018, patient around 900 which is 8.9% were new patients received hemodialysis. The prevalence of people living with ESKD and treatment with hemodialysis has been increasing each year. Nearly a haft of hemodialysis patients in Cambodia (47%) receives hemodialysis treatment twice a week and other patients receive irregular hemodialysis. As a result, many patients in Cambodia are unable to adhere the recommended guideline. Additionally, around 90 % patients experience complication before and during hemodialysis session such as fluid overload, weakness, pale, and hypertension, according to a report from Siem Reap Provincial Referral Hospital 2023.

Patient education is a process that empowers patients, and their families to learn about health conditions, treatment options, and self-management strategies. Self-management is a critical approach for patients undergoing hemodialysis. Effective patient education can enhance patients' understanding of their condition, empower them to engage in behaviors that promote self-management, and reduce complications before, during and after hemodialysis treatment.

This study aims to develop and evaluate the efficacy of a self-management program focused on improving the knowledge and self-management behaviors of hemodialysis patients at Siem Reap Provincial Referral Hospital, Cambodia. By providing targeted education on basic of disease, basic of hemodialysis, its complication, reading laboratory data, medication adherence and daily care.

This study will use a quasi-experimental pre- and post-design to improve in patients' knowledge and self-management behavior for CKD patients maintaining on hemodialysis.

The study will be conducted at Siem Reap Provincial Referral Hospital, Cambodia. The study population consists of patients undergoing hemodialysis in this hospital, who meet the criteria. The written informed consent will be taken from patients.

Convenience sampling will be employed to recruit participants, with patients selected based on their availability and willingness to take part in the study. All eligible patients who meet the inclusion criteria will be invited to participate. The sample size was calculated by using the G*Power 3.1.9.7 software, on the basis effect size of 0.5, an estimated power of 0.8, and of 0.05. A two tailed test was used to calculate that the sample should be 34 patients. However, because of this pilot nature, we include all patients who meet the inclusion criteria (n= 54).

Data analysis will be performed using statistical software SPSS. A descriptive and inferential statistical analysis will be used to address the research objectives. Descriptive statistics will summarize baseline sociodemographic and clinical history. All data will be counted and distribution, mean and standard deviation (SD) will be calculated. Reliability will be tested using Cronbach's alpha on both the self-management questionnaire and the knowledge questionnaire. Factor analysis will also be conducted on the self-management questionnaire. The results of each questionnaire at each point will be examined for mean, SD, and normality. Paired t-test will use to compare the different mean score of self-management, knowledge, QoL, self-monitoring, and physical and laboratory data at baseline and endline. One-way repeated ANOVA or Friedman's test after checking the normality on self-monitoring and physical and laboratory data. Relations among knowledge, self-management behavior, self-monitoring, physical and laboratory data, and QoL will be assessed by regression analysis and correlations. Qualitative data will be transcribed, coded, and categorized for understanding patient's experience and chanted. Statistical significance will be set as < 0.05.

Through participation in this study, hemodialysis patients will develop comprehensive knowledge, enhancing their self-management behaviors, and empowering them to manage their condition independently. The statistically significant result of this study can be provided a foundation for the development of education programs across Cambodia, ultimately improving the QOL for CKD patients undergoing hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older.
* Patients receive hemodialysis treatment at least once a week, irrespective of gender, causes of introduction of dialysis, and number of years since dialysis was introduced.

Exclusion Criteria:

* Patients with psychiatric disorders or cognitive impairments diagnosed by the medical doctor that may hinder their ability to participate in the educational sessions and self-management.
* Patients don't have shunt.
* Patients receiving additional dialysis treatment such as peritoneal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Patients' self-management behavior | 3 months after baseline data collection
  Patients' self-management behavior, as measured by the researcher-developed questionnaire. The questionnaire has 20 items with the 4 Likert scale (3: applies to me very much, 2: applies to me to a considerable degree, 1: applies to me to some degree, 0: does not apply to me). Score rang is from 0 to 60.

SECONDARY OUTCOMES:
Patient' knowledge | 3 months after baseline data collection
  Patients' knowledge score, measured by the questionnaire developed by the research team (the same as the 1)) based on our educational booklet. The questionnaire has 25 items with "True", "False", and "Don't know" answers. True = 1 point, and "False" and "Don't know" = 0 point. Score range is from 0 to 25. The research team also input 3 additional questions include 3 examples of good protein-contain food, 3 example of rich in carbohydrate food, and 3 example of high potassium fruits.
Quality of Life Measurement Using the EQ-5D-5L: A Five-Dimensional Assessment of Health Status | 3 months after baseline data collection
  Quality of life: measured by the 5-level EQ-5D version (EQ-5D-5L) was introduced by the EuroQoL group in 2009, and Khmer version was developed in 2011. The EQ-5D-5L have five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state
Self-monitoring | 3 months after baseline data collection
  Self-monitoring: the data will be extracted from the patient self-monitoring notebook. Count the number of days in a month (30 or 31 days) that each self-care behavior was implemented and divide by the number of days in a month to produce a percentage. Baseline data will be calculated based on the implementation status in the month of consent.
Blood pressure data | 3 months after baseline data collection
  Blood pressure (in millimeters of mercury) is measured by the nurse when the patient arrives for dialysis. The average of blood pressure at the start of dialysis on the day of dialysis for that month (one month) will be calculated.
Weight data | 3 months after baseline data collection
  Weight (in kilograms) is measured by the nurse when the patient arrives for dialysis. The average of weight at the start of dialysis on the day of dialysis for that month (one month) will be calculated.
Creatinine data | 3 months after baseline data collection
  Creatinine level is collected from laboratory data in the patient record at both baseline and endline.
Urea data | 3 months after baseline data collection
  Urea level is collected from laboratory data in the patient record at both baseline and endline.
Qualitative data | 3 months after baseline data collection
  Qualitative data Once a month (preferably during the last week of dialysis), the nurse conducts an unstructured interview at the bedside with the patient on dialysis about his/her experiences and changes after participating in the program. Patients are free to describe their experiences and changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Siem Reap Provencal Referral hospital, Siem Reap, Siem Reap, Cambodia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lightfoot CJ, Nair D, Bennett PN, Smith AC, Griffin AD, Warren M, Wilkinson TJ. Patient Activation: The Cornerstone of Effective Self-Management in Chronic Kidney Disease? Kidney Dial. 2022 Mar;2(1):91-105. doi: 10.3390/kidneydial2010012. Epub 2022 Mar 3. PMID 37101653
- [Background] Weir MR. Hypervolemia and blood pressure: powerful indicators of increased mortality among hemodialysis patients. Hypertension. 2010 Sep;56(3):341-3. doi: 10.1161/HYPERTENSIONAHA.110.156588. Epub 2010 Jul 12. No abstract available. PMID 20625072
- [Background] Lawless MT, Tieu M, Feo R, Kitson AL. Theories of self-care and self-management of long-term conditions by community-dwelling older adults: A systematic review and meta-ethnography. Soc Sci Med. 2021 Oct;287:114393. doi: 10.1016/j.socscimed.2021.114393. Epub 2021 Sep 10. PMID 34534780
- [Background] Thomas B, van Pelt M, Mehrotra R, Robinson-Cohen C, LoGerfo J. An estimation of the prevalence and progression of chronic kidney disease in a rural diabetic cambodian population. PLoS One. 2014 Jan 22;9(1):e86123. doi: 10.1371/journal.pone.0086123. eCollection 2014. PMID 24465909